CLINICAL TRIAL: NCT06707766
Title: Comparison of Oculomotor Exercises and Muscle Energy Technique on Visual Fatigue Among Patients Having Forward Head Posture
Brief Title: Comparison of Oculomotor Exercises Versus Suboccipital METs on Visual Fatigue Among FHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/02020 Amna Rashid.
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Forward Head Posture; Visual Fatigue
Keywords: forward head posture; visual fatigue; Craniovertebral angle; proprioception; suboccipital muscles; , oculomotor exercises; muscle energy technique (PIR; VOR(vestibulo- ocular reflex); cervical spine.
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oculomotor exercises along with conventional therapy (Experimental): oculomotor exercises along with conventional therapy
  Interventions: Other: Oculomotor Exercise along with conventional Therapy
- sub-occipital muscle energy technique along with Conventional Therapy (Experimental): Sub-occipital muscle energy technique (PIR) 3 reps * 1 set conventional therapy: Hot pack 20 minutes
  Kendall exercises were performed as follows:
  strengthening exercise: 12 repetitions* 3 sets, 2-8 sec hold stretching exercise was: 3 reps* 30 seconds' hold
  1. Strengthening the deep cervical flexors
  2. Stretching the cervical extensors
  3. Strengthening shoulder retraction
  4. Stretching of the pectoralis major muscle
  Interventions: Other: sub-occipital muscle energy technique along with Conventional Therapy

INTERVENTIONS:
Other: Oculomotor Exercise along with conventional Therapy — Oculomotor Exercises: Saccadic eye movement, Smooth pursuit, Adaptation X1, Adaptation X2.
  Time duration will be 2 minutes for each exercise.
  conventional therapy: hot pack 20 mins Kendall exercises: Strengthening the deep cervical flexor, Stretching the cervical extensors, Strengthening shoulder retraction, Stretching of the pectoralis major muscle strengthening exercise: 12 repetitions* 3 sets, 2-8 sec hold stretching exercise was: 3 reps* 30 seconds' hold
  Total duration of treatment would be 4 weeks, 3 days a week with total 12 sessions.
  Arms: oculomotor exercises along with conventional therapy
Other: sub-occipital muscle energy technique along with Conventional Therapy — Sub-occipital muscle energy technique (PIR) 3 rep * 1 set with 20 sec hold
  conventional therapy: hot pack 20 mins Kendall exercises: Strengthening the deep cervical flexor, Stretching the cervical extensors, Strengthening shoulder retraction, Stretching of the pectoralis major muscle
  strengthening exercise: 12 repetitions* 3 sets, 2-8 sec hold stretching exercise was: 3 reps* 30 seconds' hold
  Total duration of treatment would be 4 weeks, 3 days a week with total 12 sessions.
  Arms: sub-occipital muscle energy technique along with Conventional Therapy

SUMMARY:
The aim of this research is to compare the effect of Oculomotor Exercises and Muscle energy technique on visual fatigue, proprioception, Craniovertebral angle among patients having Forward head posture.. It will raise awareness about the link between posture and visual health, encouraging early identification of visual symptoms associated with FHP, enhance recovery outcomes, improve functional performance, and promote a holistic treatment approach, ultimately provide benefit to population.

DETAILED DESCRIPTION:
Studies have shown that integrating eye exercises with neck strengthening exercises has a significant effect in managing symptoms associated with visual disturbances and neck pain. For instance, a study conducted in 2024 to investigate the effect of oculomotor exercises in patients having chronic neck pain. Based on the result, they found that incorporating oculomotor exercises along with conventional exercises into treatment plan can significantly improve gaze stability, proprioception, visual acuity and fatigue in chronic neck pain patients. In 2023 study investigate the effectiveness of manual techniques for the management of FHP. They found that sub-occipital muscle energy technique is effective in improving CVA, cervical range of motion and postural alignment. study conducted in 2023 investigated the comparative effect sub-occipital muscle energy technique vs sub-occipital release in mechanical neck pain and FHP population. They concluded that group receiving MET show significant improvement in CVA, NDI and Cervical ROMs. Another research concluded that Sub-occipital muscle energy technique incorporating with proprioceptive training are effective in improving joint position sense (proprioception) and CVA in FHP population. A study evaluate the effectiveness of eye exercises on computer vision syndrome. They concluded the ocular exercises are effective in reducing visual fatigue symptoms such as eye itching, dryness and headache.

This research is innovative as it explores the interconnected roles of ocular muscles and sub-occipital muscles on visual fatigue, proprioception, and postural imbalances, particularly in FHP patients. As Literature suggest that tightness of suboccipital affect somatosensory input and proprioceptive information crucial for head and eye coordination. Thus, offering a comprehensive view of how FHP and visual fatigue are interconnected. Furthermore, the integration of oculomotor exercises in managing FHP-related visual fatigue is an underexplored as the existing literature primarily focuses on the musculoskeletal consequences of forward head posture and ocular exercises for visual disturbance without exploring the interaction between these factors. This research aimed to bridge the existing gap in literature by providing evidence-based guidance on the effectiveness of METs and oculomotor exercises in the management of visual symptoms associated FHP.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years
* Both Male and Female
* Diagnosed patients of Forward head posture, Craniovertebral Angle less than 50 degree.
* Patients having Asthenopia survey questionnaire (ASQ-17) score of 13 or higher.

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.
* Pre-existing medical conditions that cause visual issues such as conjunctivitis, cataract, Strabismus anomaly, glaucoma and those undergoing any eye treatment.
* Any previous neck and Eye surgery.
* Cervical conditions such as cervical radiculopathy, non-specific neck pain, and TMJ dysfunction that cause visual disturbances.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
visual fatigue | 4 weeks
  ; Visul fatigue can be assessed by using Asthenopia Survey Questionnaire (ASQ-17). Responses are marked using four-point Likert scale with total score 51. Score range from 0-13 indicates no asthenopia, whereas the score range between 13-51 indicate asthenopia and need medical attention
propioception | 4 weeks
  cervical proprioception can be assed Cervical Joint Position Error (JPE) Test. Values > 4.5 degree indicate proprioception deficit
Craniovertebral Angle | 4 weeks
  Craniovertebral Angle can be measured by usng ON PROTRACTOR google App. Craniovertebral angle (CVA) values for individuals with moderate-severe forward head posture ranged from 40.7° to 43.2°, and for those with mild FHP, values ranged from 46.9° to 49.1 FHP. However, angle between 50- 57 degree is consider as normal.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aneela Zia, ms-ompt, Principal Investigator — Riphah International University
Locations (3):
- Pakistan (3):
  - Capital Diagnostic Center Islamabad, Islamabad
  - Care plus Medical Center, Islamabad
  - National Institute of Rehabilitation, Islamabad

IPD SHARING:
Plan to Share IPD: No